CLINICAL TRIAL: NCT02617017
Title: Buspirone Treatment of Iatrogenic Dyskinesias in Advanced Parkinson' Disease. Multicenter, International, Placebo-controlled, Randomised, Double Blind Trial
Brief Title: Buspirone Treatment of Iatrogenic Dyskinesias in Advanced Parkinson' Disease
Acronym: BUSPARK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P130909; 2015-002332-41 (EudraCT Number)
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Parkinson
Keywords: Parkinson disease; Levodopa induce dyskinesia
MeSH Terms: conditions — Parkinson Disease | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buspirone (Experimental)
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — Capsules of buspirone will be administered orally once a day for 2 weeks (10mg, morning), BID for 2 further weeks (20 mg, morning and evening), TID between weeks 5 and 12 (third intake at noon)
  Arms: Buspirone
Drug: Placebo — Capsules of placebo will be administered orally once a day for 2 weeks (10mg, morning), BID for 2 further weeks (20 mg, morning and evening), TID between weeks 5 and 12 (third intake at noon)
  Arms: Placebo

SUMMARY:
Parkinson's disease (PD) is one of the most common neurodegenerative diseases, with a higher prevalence in the elderly. Levodopa induced dyskinesias (LID) are a major motor complications that impair quality of life for patients with PD. The mechanisms of these dyskinesias remain unclear, but several hypotheses have been put forward: non continuous, pulsatile stimulation of dopaminergic receptors, or alterations of other neurotransmitters within the motor striatum such as glutamate and serotonin.

Few strategies are now available to treat severe LID:

* Medications: reduction of dopaminergic treatment, addition of amantadine,
* Functional neurosurgery. The purpose of this study is to investigate the efficacy of buspirone in PD patients suffering from dyskinesias. The role of serotonin in the occurrence of LID was recently demonstrated in transplant PD patients and a test double-blind, single dose was achieved. Following administration of 10 mg oral buspirone, a 5HT1A agonist, LID were clearly improved. A antidyskinetic effect of buspirone had already been reported in 1991 and 1994, but identification of buspirone as a serotonin receptor agonist has been reported more recently.

This trial is aimed at (1) validate the serotoninergic hypothesis of hyperkinetic levodopa induced dyskinesias (LID) in Pakinson's disease patients, (2) evaluate, in a phase 3 trial, the motor efficacy of buspirone to improve LID vs placebo, (3) look at a possible dose/effect relationship and (4) check the hypothesis of a better therapeutic ratio using the association of buspirone and amantadine instead than a single drug.

ELIGIBILITY:
Inclusion Criteria

* The subject is an out-patient between 35 year and 80 years of age
* Diagnosis of idiopathic Parkinson's disease according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnosis Criteria
* Dyskinesias are present more than 25% of the waking day according to item 4-1 of MDS-UPDRS
* Dyskinesias are at least moderately disabling item 4-2 of MDS-UPDRS replaced by Dyskinesias are at least slightly disabling item 4-2 of MDS-UPDRS (amendment n°2)
* The subject is able to identify dyskinesia, ON and OFF, and apply to his/her own state
* Stable dose of anti-Parkinsonian drugs for at least 4 weeks up to the screening
* The subject is considered as being optimally treated at the time of inclusion
* Written and signed informed consent to participate in the study
* Maximal Hoehn and Yahr staging : III in "ON" phases, IV in "OFF"
* Active affiliation to social security
* Menopausal or under contraception for woman

Exclusion Criteria

* Female subjects : pregnant or lactating
* Atypical parkinsonian syndrome
* Weight less than 40 Kgs
* Mini-Mental State Examination (MMSE) less than 24
* The subject is participating in another clinical study within the past 12 weeks
* Planned participation in another therapeutic clinical study
* Previous treatment with buspirone, less than 6 months before Week 0
* Known allergy to buspirone
* Known lactose intolerance
* Clinically significant illness that might interfere with the study
* Dementia or other psychiatric illness
* Drug or alcohol abuse replaced by Substance use disorder (alcohol i.e. > 3 drinks per day for men and > 2 drinks per day for women,drug, medicinal product) (amendment n°1)
* Legal incapacity or limited legal capacity
* Deep brain stimulation performed less than 12 months before protocol initiation, or unstable parameters of stimulation 4 weeks before week 0
* Severe renal and / or hepatic impairment
* History of seizures or epilepsy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Between-group comparison of changes in UDysRS scores | Between baseline and week 12

SECONDARY OUTCOMES:
Comparison, in both groups of patients of Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part 3-4 (efficacy) | At week 0,Week2, Week4, Week12, Week13
Comparison, in both groups of patients of MDS-UPDRS part 1-2 (quality of life) | At week Week-2, Week0, Week2, Week4, Week12, Week13
Comparison, in both groups of patients of PDQ-39 (quality of life) | At week 0 and week 12
Comparison, in both groups of patients of side effects (tolerance) | At week Week-2, Week0, Week2, Week4, Week12, Week13
Maximum dose accepted by patients (tolerance) | At week Week-2, Week0, Week2, Week4, Week12, Week13

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rémy, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWNED BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217